CLINICAL TRIAL: NCT01372319
Title: Assessment of Advanced Glaucomatous Visual Field Loss and Its Impact on Visual Exploration, Activities of Daily Living (ADL) and Quality of Life (QoL)
Acronym: GlaucomaEXPLOR
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Professor Dr. med Ulrich Schiefer, University Hospital Tuebingen
Other Study IDs: 085/2011B02
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: glaucoma; binocular visual field loss; semi-automated kinetic perimetry (SKP); quality of life (QoL); visual exploration; on-road car driving; driving simulator
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma Patients (OAG, Aulhorn stages II - IV): Manifest glaucoma (OAG, Aulhorn stages II - IV) with advanced binocular visual loss, as obtained by semi-automated kinetic perimetry (SKP), no study medication
- Normal subjects: male+female > 18 years

SUMMARY:
The purpose of this explorative study, targeting subjects with advanced binocular glaucomatous visual field loss, is: (i) to identify the perimetric / psychophysical method, that is most closely correlated with an individually assessed quality of life (QoL) score, using a validated questionnaire (NEI-VFQ 25), (ii) to determine, whether gaze-related (exploratory eye movements) or visual field-related (eyes steadily fixating) OR attention-related parameters are better for the characterization of the visual capacities that are necessary for activities of daily living (ADL), as represented (iia) by a standardized visual search task and (iib) by an on-road car driving feasibility study.

Further this study is intended to introduce and analyse a novel diagnostic method for recording and evaluating exploratory eye movements (gaze-related perimetry) in a clinical setting. A similar procedure has recently been introduced by Murray et al. However, their set-up is based on a video monitor and, therefore, restricted to the central visual field (eccentricity < 25°) and limited with regard to the dynamic range of the stimulus luminance. Since our new gaze-related perimetry is designed to be implemented in a conventional cupola perimeter, it should be widely available as a potent diagnostic tool, for screening purposes, or for clinical surveys by general ophthalmologists or clinical research groups.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma subjects Primary inclusion criteria: Open angle glaucoma (OAG), according to the classification of the European Glaucoma Society (EGS)11 with advanced binocular visual loss (i.e stages II - IV according to the classification after Aulhorn et al.4, as obtained by semi-automated kinetic perimetry (SKP) or automated static threshold-related, slightly supraliminal perimetry (sAS) 3,10 22 [Grid 30°-NO (192 test points), stimulus Goldmann size III = 26´, OCTOPUS 101/900 perimeter (Haag-Streit Inc., Köniz, Switzerland)].
* Further inclusion criteria: (i) General: physical, intellectual and linguistic abilities, necessary to understand the test requirements: no mobility limitations, Minimental Status Examination Test score above 24, adequate knowledge of the German language, willingness to comply with the protocol, > 18 years, informed consent.

(ii) Ophthalmological: spherical ametropia max. ± 8 dpt, cylindrical ametropia max. ± 3 dpt, distant visual acuity > 10/20, isocoria, pupil diameter > 3 mm.

- Normal subjects (i) General inclusion criteria: Physical, intellectual and linguistic abilities needed to understand the test requirements: no mobility limitations, Minimental Status Examination Test score above 24, adequate knowledge of the German language, willingness to comply with the protocol, > 18 years, informed consent.

(ii) Ophthalmological inclusion criteria: maximum allowed spherical ametropia at distance is ± 6.00 diopters and the maximum cylindrical ametropia is ± 2 dpt. The best corrected distance visual acuities are ≥ 20/20 (1.0) for those aged up to 60 years; > 20/25 (0.8) for those aged between 60 and 70 years; ≥ 20/33 (0.6) for those aged more than 70 years. All participants manifest equal pupil size, pupil diameter > 3 mm, no relative afferent pupillary defect, intraocular pressure ≤ 21 mmHg, normal anterior segments, no clinically relevant media opacities, normal appearance of the optic disc (cup to disc ratio = CDR ≤ 0.5, intraocular difference of CDR < 0.3) and normal central and peripheral fundus findings on direct and indirect undilated ophthalmoscopic examination.

Exclusion Criteria:

* Glaucoma subjects (i) General exclusion criteria: pregnancy, nursing, asthma, HIV+ or AIDS, history of epilepsy or significant psychiatric disease, history of drug and alcohol abuse, Minimental Status Examination Test score below 24, medications known to affect visual field sensitivity.

(ii) Ophthalmological exclusion criteria: diabetic retinopathy, infections (e.g. keratitis, conjunctivitis, uveitis), severe dry eyes, miotic drug, amblyopia, squint, nystagmus, albinism, any ocular pathology, in either eye, that may interfere with the ability to obtain visual fields, disc imaging or accurate IOP readings, keratoconus, intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening, history or signs of any visual pathway affection other than glaucoma, allergies with regard to topic glaucoma medication, history or presence of macular disease and / or macular edema, ocular trauma.

- Normal subjects

(i) General exclusion criteria: mental or neurological diseases, diabetes mellitus, history of coronary heart disease, stroke, migraine, vasospasm / Raynaud's disease; drugs indicating severe systemic diseases (e.g. anti-diabetic or anti-hypertensive medication for subjects under 70 years of age), drugs or medications influencing reaction time, pregnancy, nursing; history of drug and alcohol abuse. Subjects over 70 years of age will not be excluded for use of anti-hypertensive medication.

(ii) Ophthalmological exclusion criteria: Amblyopia, strabismus, ocular motility disorders, retinal pathology, glaucoma, suspicion of glaucoma, ocular hypertension or any other sign of other optic neuropathy, macular degeneration, pathological color vision test results (Ishihara Standard Pseudoisochromatic Plates), eye surgery (except cataract surgery), any type of refractive surgery; history or signs of neuro-ophthalmological diseases, acute infections, diabetic retinopathy, use of miotic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First year: 10 glaucoma patients, with advanced binocular visual loss and 10 age-related (+ 5 years of age) and gender-matched normal subjects. Second year: Extension to a total number 30 glaucoma patients, with advanced binocular visual loss and 30 age-related (+ 5 years of age) and gender-matched normal subjects (according to the sample size estimation), if additional budget available.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Identification of the perimetric / psychophysical method, that is most closely correlated with an individually assessed quality of life (QoL) score. | 2 years
  Quality of life (QoL), assessed with the NEI-VFQ 25 questionnaire, is better correlated with the modified ESTERMAN score, based on the binocular semi-automated kinetic perimetry of the 90° visual field (90° SKP) than with the number of affected test locations (local sensitivity < 10 dB) according to the binocular integrated visual field (IVF).
Determination of the most appropriate parameters (gaze-related ; visual field-related; attention-related) for the characterization of the visual capacities for activities of daily living | 2 years
  Performance regarding activities of daily living (ADL), as represented by the "supermarket special offer search task", are better correlated with (the modified ESTERMAN score, based on) the intact binocular gaze field than with (the modified ESTERMAN score, based on) the binocular semi-automated kinetic perimetry of the 90° visual field (90° SKP) OR the with the number of affected test locations (local sensitivity < 10 dB) of the binocular integrated visual field (IVF) OR the UFOV risk score.

SECONDARY OUTCOMES:
Comparison of the comprehensive psychophysical examinations | 2 years
  The scotoma extent, assessed with MAFOV, is equal to the scotoma extent assessed with the fast thresholding conventional static automated perimetry (SAP) (GATE strategy, Grid 30-S). Additionally, test/re-test reliability will be assessed with regard to (i) MAFOV and (ii) SAP (as described above), assuming that test/retest reliability is identical between MAFOV and SAP.
Comparison and evaluation of two different assessments of visual exploration under real-life scenarios ("supermarket special offer search task", "on-road car driving" by means of a dual brake vehicle (optional: driving simulator) | 2 years
  Performance regarding acitivities of daily living (ADL), as assessed by the "supermarket special offer search task" and the "on-road car driving pilot study", are better correlated with (the ESTERMAN score, based on) the intact binocular gaze field than with (the ESTERMAN score, based on) the binocular semi-automated kinetic perimetry of the 90° visual field (90° SKP) OR the with the number of affected test locations (local sensitivity < 10 dB) of the binocular integrated visual field (IVF) OR the UFOV risk score.
Descriptive assessment of structure-function relationships by comparing the results of the different perimetric tests with the morphometric results of HRT III | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr.med., Principal Investigator — Centre for Ophthalmology Institute for Ophthalmic Research University of Tübingen
Locations (1):
- Centre for Ophthalmology University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Kasneci E, Sippel K, Aehling K, Heister M, Rosenstiel W, Schiefer U, Papageorgiou E. Driving with binocular visual field loss? A study on a supervised on-road parcours with simultaneous eye and head tracking. PLoS One. 2014 Feb 11;9(2):e87470. doi: 10.1371/journal.pone.0087470. eCollection 2014. PMID 24523869
- [Background] Kübler T, Kasneci E, Rosenstiel W, Schiefer U, Nagel K, Papageorgiou E. Stress-indicators and exploratory gaze for the analysis of hazard perception in patients with visual field loss. Science Direct, Transportation Research Part F 24: 231-43, 2014
- [Derived] Kasneci E, Sippel K, Heister M, Aehling K, Rosenstiel W, Schiefer U, Papageorgiou E. Homonymous Visual Field Loss and Its Impact on Visual Exploration: A Supermarket Study. Transl Vis Sci Technol. 2014 Nov 3;3(6):2. doi: 10.1167/tvst.3.6.2. eCollection 2014 Oct. PMID 25374771
- [Derived] Sippel K, Kasneci E, Aehling K, Heister M, Rosenstiel W, Schiefer U, Papageorgiou E. Binocular glaucomatous visual field loss and its impact on visual exploration--a supermarket study. PLoS One. 2014 Aug 27;9(8):e106089. doi: 10.1371/journal.pone.0106089. eCollection 2014. PMID 25162522